CLINICAL TRIAL: NCT03212664
Title: Effectiveness of Physical Therapy Exercises in Hyperkyphosis
Brief Title: Physical Therapy Exercises in Hyperkyphosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Scottish Rite Hospital for Children (Other)
Responsible Party: Principal Investigator, Karina Zapata, PT, DPT, PhD, research therapist, Texas Scottish Rite Hospital for Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1143
Record Dates: First submitted 2017-07-03; First posted 2017-07-11 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Hyperkyphosis
MeSH Terms: conditions — Kyphosis | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Other): Schroth-based physical therapy exercises for patients who agree to participate in exercises. Will be compared to observation-only treatment
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — physical therapy exercises

SUMMARY:
This proposal is a single center preliminary prospective cohort trial that evaluates patients with hyperkyphosis. Participants will receive physical therapy exercises and be followed for the above outcome measures over time. The treatment arm will receive training in one-time training in kyphosis-specific exercises.

It is hypothesized that participants receive physical therapy exercises will demonstrate improved outcome measures over time. Also, it is hypothesized that participants who receive kyphosis-specific exercises will demonstrate significantly improved perceived quality-of-life and significantly reduced pain, compared to participants who receive generalized back exercises after 6 months.

Also, it is hypothesized that a kyphosis-specific SAQ will demonstrate satisfactory test-retest reliability and concurrent validity.

DETAILED DESCRIPTION:
A total of 50 patients will be recruited for this study. 28 patients will be recruited for both groups, or 14 participants per group. Patients will be randomized by an independent research assistant who will draw the group number from a hat. We assume less than 15% attrition, which results in 12 participants per group.

Patients in both groups will ideally be followed after 6 months, unless the patient's treating orthopaedic surgeon schedules them for a visit up until 12 months later.

Group 1(Kyphosis-specific exercise Group): Patients will receive a one-time treatment consisting of kyphosis-specific exercises that promote depressing the thoracic convexity.

Group 2 (Generalized exercise group): Patients will receive a one-time treatment consisting of core strengthening, hamstring stretching, and generalized back extension exercises.

Patients in each group will be asked to perform these exercises at home about 10 minutes a day, 3 times a week.

Each patient will be given access to a software application though PT PAL on their smart phone (or computer). Patients will be asked to use the app whenever they perform their exercises throughout the 6 month period. Patients must turn off the app after 15 minutes for the app to count the exercise session as complete. Each physical therapist participating in the study will have administrator access to monitor exercise adherence for their respective patients at any time as a tool to maximize exercise adherence.

Each patient will also be asked about their pain intensity on a monthly basis through a secure database (REDCap).

5. Study Procedures: Group 1 or 2

Month 0 (40 minutes):

* X-ray of back [standard of care]
* Picture of back [research]
* Physical therapy program [research]
* Two surveys on how kyphosis affects the patient [research]
* Physical examination [research]

Week 2 (10 minutes):

* Two surveys at home on how kyphosis affects the patient [research]

Months 1-5 (2 minutes)

• Monthly survey at home regarding your back pain [research]

Month 6-12 (40 minutes):

* X-ray of back [standard of care]
* Picture of back [research]
* Two surveys on how kyphosis affects the patient [research]
* Physical examination [research]

These x-rays will not need to be ordered as a study procedure.

5a. Sub-Study: Aim 2 Kyphosis-Specific SAQ (K-SAQ) The secondary aim of this study is to assess the psychometric properties of a kyphosis-specific SAQ and evaluate the test-retest reliability and concurrent validity of this kyphosis-specific SAQ.

The original study design included enrolling a total of 28 patients, all of whom would receive and complete the SRS-22 and the kyphosis-specific SAQ at baseline, two weeks, and 6-12 month follow-up.

At the conclusion of initial enrollment, 21 patients had been enrolled and six (6) were lost to follow-up. Of the 21 total patients, 15 completed Aim 1 of this study, not all of which completed Aim 2.

During analysis, we found statistical significance for the test-retest reliability and concurrent validity of the K-SAQ, but due to weak enrollment and completion of the questionnaires at baseline and two weeks, we are enrolling more patients for Aim 2 of the original study design and will end enrollment for Aim 2 at the conclusion of 25 completed responses of the K-SAQ and SRS-22 for both baseline and 2-week follow-up.

We will increase enrollment from 28 patients to 50 patients.

Patients in this sub-group must be diagnosed with hyperkyphosis, have a Cobb angle of at least 50°, and be 8-21 years old. Exclusion criteria includes: scoliosis greater than 25°, current brace wear, and previous spine surgery. Specific treatment is not a part of this sub-group.

Patients enrolled in the Kyphosis-specific SAQ Sub-group of the PPKS Registry (STU 032011-130) will be included within this sub-group for data analysis.

6. Criteria for Inclusion of Subjects: Patients with a diagnosis of hyperkyphosis meeting the following inclusion criteria will be eligible to participate: ages 10 to 18 years, Cobb angles at least 50°, and pain >2 on the VAS during the past week.

7. Criteria for Exclusion of Subjects:

Patients will be excluded according to the following exclusion criteria:

scoliosis greater than 25°, conditions preventing understanding and compliance with an exercise schedule, current brace wear, previous spine surgery, inability to commit to at least 15 minutes of exercises for 3 days a week, and pain <2 on the VAS during the past week.

8. Sources of Research Material: Baseline participant characteristics will include age, sex, ethnicity, Risser sign, height, weight, BMI, curve magnitude of a lateral radiograph, and location of the kyphosis apex. The lateral radiograph information will be obtained from Synapse, a radiology information system at TSRH.

Exercise adherence will be recorded including the length of exercise sessions and total duration of PT until the patient is discharged to a HEP. HEP adherence will be calculated as the percentage of prescribed exercises completed from baseline to 6 months.

9. Recruitment Methods and Consenting Process: Patients will be screened by the investigators, participating physical therapists, or research coordinator to determine whether inclusion criteria is met. If the patient is eligible for this trial, the patient will be offered enrollment to the patient and caregiver. Appropriate patient assent and caregiver consent to participate in the trial will be obtained per IRB protocol. The patient will then choose to be in either the treatment or observation group.

10. Potential Risks: Identifiable risk associated with participation in this study would be a potential loss of confidentiality and tired or sore muscles from the exercises.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of hyperkyphosis
* ages 10 to 18 years
* Cobb angles at least 50°
* pain >2 on the VAS during the past week.

Exclusion Criteria:

* scoliosis greater than 25°
* conditions preventing understanding and compliance with an exercise schedule
* current brace wear
* previous spine surgery
* inability to commit to at least 15 minutes of exercises for 3 days a week
* pain <2 on the VAS during the past week.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2014-08-05 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
survey | 6 month follow-up
  19 items that identify factors related to exercise adherence, app usability and acceptability

SECONDARY OUTCOMES:
pain intensity | baseline
  Numeric Pain Rating Scale
pain intensity | 6 month follow-up
  Numeric Pain Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Karina A Zapata, PhD, Principal Investigator — Texas Scottish Rite Hospital for Children
Locations (1):
- Texas Scottish Rite Hospital for Children, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zapata KA, Wang-Price SS, Fletcher TS, Johnston CE. Factors influencing adherence to an app-based exercise program in adolescents with painful hyperkyphosis. Scoliosis Spinal Disord. 2018 Jul 18;13:11. doi: 10.1186/s13013-018-0159-x. eCollection 2018. PMID 30027121